CLINICAL TRIAL: NCT01510184
Title: A Phase 3, Open-label, Multicenter, Randomized Study of Sequential Zevalin (Ibritumomab Tiuxetan) Versus Observation in Patients at Least 60 Years of Age With Newly Diagnosed Diffuse Large B-cell Lymphoma in PET-negative Complete Remission After R-CHOP or R-CHOP-like Therapy
Brief Title: Study of Zevalin Versus Observation in Participants at Least 60 Years Old With Newly Diagnosed Diffuse Large B-cell Lymphoma in Positron Emission Tomography (PET)-Negative Complete Remission After Rituximab-Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (R-CHOP) or R-CHOP-like Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPI-ZEV-11-301
Record Dates: First submitted 2012-01-06; First posted 2012-01-13 (Estimated); Results first posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-11

CONDITIONS: Diffuse Large B-cell Lymphoma; Follicle Center Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — ibritumomab tiuxetan; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zevalin (Experimental): Participants received rituximab 250 milligram per meter square (mg/m^2) by intravenous infusion on Day 1. If required by the governing regulatory agency, rituximab was to be followed 4 hours later by In-111-Zevalin 5.0 millicurie (mCi) on Day 1. And on Days 7-9: participants received rituximab 250 mg/m^2 by intravenous infusion, followed 4 hours later by Y-90-Zevalin 0.4 millicurie/kilogram (mCi/kg) 10-minute intravenous push (0.3 mCi/kg in participants with a platelet count in 100,000/ microliter [μL] to 149,000/μL).
  Interventions: Drug: Zevalin; Drug: Y-90-Zevalin; Drug: Rituximab; Drug: In-111 Zevalin
- Observation (No Intervention): Participants who were randomized in this arm group did not receive any anti-lymphoma therapy unless they had a relapse of their disease.

INTERVENTIONS:
Drug: Zevalin — Zevalin administered intravenous infusion.
  Other Names: Ibritumomab Tiuxetan
  Arms: Zevalin
Drug: Y-90-Zevalin — Y-90-Zevalin administered by intravenous infusion.
  Arms: Zevalin
Drug: Rituximab — Rituximab administered by intravenous infusion.
  Arms: Zevalin
Drug: In-111 Zevalin — In-111-Zevalin administered by intravenously.
  Arms: Zevalin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Zevalin compared with observation alone in participants who are in PET-negative complete remission after first-line R-CHOP or R-CHOP like therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participant was 60-years of age or older at time of randomization
2. Histologically confirmed Ann Arbor stage II, III, or IV diffuse large B-cell lymphoma (DLBCL); or follicular lymphoma (FCL) Grade 3B according to the Revised European American lymphoma (REAL)/ World health organization (WHO) classification (from initial diagnosis made prior to starting R-CHOP therapy. Results from a pre R-CHOP marrow shall be available for review.
3. Local pathology review confirming the DLBCL diagnosis and cluster of differentiation 20 (CD20) positivity, and no evidence of DLBCL in bone marrow upon confirmation of complete remission (CR).
4. A paraffin block or original slides available for confirmatory pathology review. Participants may be randomized based on the local pathology result.
5. Age-adjusted international prognostic index (IPI) of 1, 2, or 3. The age-adjusted IPI was defined by one point for Lactate dehydrogenase (LDH) > upper limit of normal (ULN); Stage III or IV; and Karnofsky performance status <80% or WHO/ eastern cooperative operations group (ECOG) performance status >1.
6. First-line treatment of DLBCL must have been 6 cycles of standard R-CHOP21, R-CHOP14 or dose-adjusted etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (DA-EPOCH-R) chemotherapy. Participants who received pre-phase therapy for the purpose of improving performance status prior to initiating R-CHOP are eligible.
7. Complete remission (CR) according to the International Workshop Response Criteria for non-Hodgkin's lymphoma (NHL) described by Cheson et al after first-line treatment. Computerized tomography (CT) scans of chest, abdomen, pelvis, and neck (if applicable) must have been performed within 6 weeks after the last dose of the last course of chemotherapy. Applicability of the neck CT means that the participant had involvement of the neck region by palpation / physical examination at first diagnosis.
8. A negative Fluorine-18-deoxyglucose positron emission tomography (FDG-PET) scan confirming complete response, with negative defined as a score of 1-3 on the Deauville 5-point scale used to quantify radionucleotide density in PET scans as determined locally (Morschhauser 200735).
9. Bone marrow cellularity greater than 15%, no evidence of myelodysplasia morphologically and no evidence of involvement with lymphoma either at the pre R-CHOP marrow or on repeat assessment pre-Zevalin. After completing R-chemotherapy, a repeat marrow is required for participant randomized to the Zevalin arm only.
10. A world health organization/eastern cooperative oncology group (WHO/ECOG) performance status of 0, 1 or 2.
11. Adequate hematopoietic functions: Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/ liter (L), Hemoglobin (Hgb) ≥ 9 g/dL, Platelets ≥ 100 x 10^9/L.
12. Life expectancy of 6 months or longer.
13. Written informed consent obtained according to local guidelines.

Exclusion Criteria:

1. Presence of any other malignancy or history of prior malignancy within 5 years of study entry. Within 5 years, participants treated for Stage I or II cancers are eligible provided they have a life expectancy of > 5 years. The 5-year exclusion rule does not apply to-non melanoma skin tumors and in situ cervical cancer.
2. Prior radioimmunotherapy, including radiation therapy for Non-Hodgkin's lymphoma) NHL, or any other NHL therapy.
3. Presence of primary gastric, central nervous system (CNS), or testicular lymphoma at first diagnosis.
4. Histological transformation of low-grade NHL.
5. Active hepatitis B or C.
6. Known history of human immunodeficiency virus (HIV) infection.
7. Abnormal liver function: total bilirubin > 2 × ULN unless secondary to Gilbert disease.
8. Abnormal renal function: serum creatinine > 2.0 × ULN.
9. Non-recovery from the toxic effects of chemotherapy to < grade 2, or interfering with Zevalin treatment.
10. Known hypersensitivity to murine or chimeric antibodies or proteins.
11. Granulocyte-colony stimulating factor (G-CSF) or Granulocyte macrophage-colony stimulating factor (GM-CSF) therapy within 4 weeks prior to Zevalin or observation.
12. Concurrent severe and/or medically uncontrolled disease (e.g. uncontrolled diabetes, congestive heart failure, myocardial infarction within 6 months of study, unstable and uncontrolled hypertension, chronic renal disease, or active uncontrolled infection) which could compromise participation in the study.
13. Treatment with investigational drugs less than 4 weeks prior to Zevalin or observation.
14. Major surgery less than 4 weeks prior to Zevalin or start of observation.
15. Concurrent systemic corticosteroid use for any reason except as premedication in case of known or suspected allergies to contrast media or as premedication for potential side effects of rituximab treatment. Participants on a chronic dose of prednisone for a medical condition (e.g. Asthma or autoimmune disease) less than or equal to 20 milligram (mg) daily, stable for 4 weeks, are permissible.
16. Unwillingness or inability to comply with the protocol.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-04-19 (Actual); Primary Completion 2014-10-23 (Actual); Study Completion 2014-10-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (93):
- United States (28):
  - Cancer Treatment Services Arizona, Casa Grande, Arizona
  - Sutter East Bay Hospitals, Berkeley, California
  - City of Hope, Duarte, California
  - Halifax Health Medical Center, Daytona Beach, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Piedmont Hospital Cancer Center, Atlanta, Georgia
  - St. Luke's Mountain States Tumor Institute (MSTI), Boise, Idaho
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Norton Cancer Institute, Suburban, Louisville, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Oncology Research-Park Nicollet Institute, Saint Louis Park, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Hackensack UMC / John Theurer Cancer Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Adams Cancer center, Gettysburg, Pennsylvania
  - York Cancer Center / Cancer Care Associates of York, York, Pennsylvania
  - Saint Francis Hospital, Greenville, South Carolina
  - Avera Hematology and Transplant, Sioux Falls, South Dakota
  - Associates In Oncology and Hematology, Chattanooga, Tennessee
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (5):
  - Royal Hobart Hospital, Hobart, Tasmania
  - Royal Melbourne, Parkville, Victoria
  - Royal Adelaide Hospital, Adelaide
  - Barwon Health, Geelong
  - Western Hospital, Melbourne
- Medizinische Universität Wien -AKH Wien, Vienna, Austria
- Belgium (2):
  - Nuclear Medicine Physician, Jules Bordet Institute, Brussels
  - University Hospital Gasthuisberg, Leuven
- Canada (3):
  - Thunder Bay Regional Health Sciences Centre-Regional Cancer Care, Thunder Bay, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - CSSS Champlain Charles LeMoyne, Greenfield Park, Quebec
- France (23):
  - CHU A Michallon, Grenoble, Cedex 9
  - CHU Dupuytren, Limoges, Cedex
  - CHU Amiens, Hôpital Sud, Amiens
  - CH Avignon, Avignon
  - CH de la Côte Basque, Service d'Hématologie, Bayonne
  - Hématologie - CHU Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Hopital MORVAN - CHU Brest, Brest
  - Centre François Baclesse, Comite Hématologie, Caen
  - Hôpital Henri MONDOR, Créteil
  - CHD Vendée, La Roche-sur-Yon
  - CHRU Lille- Hospital Claude Huriez, Lille
  - Institut Paoli-Calmettes, Marseille
  - CHR Metz-Thionville, Metz
  - CH de Mulhouse - Hôpital Emile Muller, Mulhouse
  - Centre Antoine Lacassagne, Nice
  - CHR Orléans, Orléans
  - Institut Curie, Paris
  - Centre Hospitalier Saint Jean, Perpignan
  - Hôpital Haut-Levêque Centre F.Magendie, Pessac
  - Centre Hospitalier René Dubos,, Pontoise
  - Service d'Hématologie Centre Henri Becquerel, Rouen
  - CHU de Brabios, Vandœuvre-lès-Nancy
- Ireland (2):
  - St James 's Hospital, Dublin
  - University Hospital Galway, Galway
- Israel (6):
  - Soroka Medical Centre, Beersheba
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Organization, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Centre, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (5):
  - Policlinico S Orsola Malpighi, Istituto di Ematologia ''L.e A. Seragnoli'', Bologna
  - New Ematologia dell'Ospedale "Spedali Civili" di Brescia, Brescia
  - Divisione di Ematoncologia, Milan
  - Azienda Ospedaliera Sant'Andrea, Roma
  - Azienda Ospedaliera San. Giovanni Battista di Torino, Dipartimento di Oncologia U.O.A Ematologia, Le Molinette,, Torino
- Netherlands (9):
  - Meander Medisch Centrum, Amersfoort
  - VU Medisch Centrum, Amsterdam
  - University Medical Centre Groningen (UMCG), Groningen
  - Spaarne Ziekenhuis, Internal Medicine/Ocology, Hoofddorp
  - Medisch Centrum Leeuwarden, Leeuwarden
  - St. Antonius Hospital, Nieuwegein
  - University Medical Center Radboud Nijmegen, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - Haga Ziekenhuis, The Hague
- Auxilio Mutuo Cancer Center, San Juan, Puerto Rico
- Spain (3):
  - Clínica Universidad de Navarra (CUN), Pamplona
  - Hospital Universitario Miguel Servet, Zaragoza
  - Miguel Servet University Hospital, Zaragoza
- United Kingdom (5):
  - Department of Haematology Bristol Royal Infirmary, Bristol
  - Poole General Hospital, Dorset
  - Beatson Cancer Centre, Glasgow
  - King's College Hospital, London
  - The Christie NHS Foundation Trust, The Christie Hospital,, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 79 participants were enrolled into the study from 19 Apr 2012 to 23 Oct 2014.
Period: Overall Study
Arm/Group | Zevalin | Observation
Started | 36 | 43
Completed | 6 | 8
Not Completed | 30 | 35
Not completed — Sponsor discretion | 28 | 28
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants classified according to the actual study treatment received, regardless of random assignment.
Groups:
- Zevalin: Participants received rituximab 250 mg/m^2 by intravenous infusion on Day 1. If required by the governing regulatory agency, rituximab was to be followed 4 hours later by In-111-Zevalin 5.0 mCi on Day 1. And on Days 7-9: participants received rituximab 250 mg/m^2 by intravenous infusion, followed 4 hours later by Y-90-Zevalin 0.4 mCi/kg 10-minute intravenous push (0.3 mCi/kg in participants with a platelet count in 100,000/μL to 149,000/μL).
- Total: Total of all reporting groups
Arm/Group | Zevalin | Observation | Total
Number analyzed (Participants) | 36 | 43 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (1.02) | 71 (1.06) | 70 (0.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 16 | 21 | 37

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) for Living Participants
Description: OS was the time from randomization to death. In living participants, survival time was censored on the last date that participants were known to be alive. OS for living participant was calculated as (end of study date/last visit date - randomization date)+ 1/30.4375. Overall Survival was summarized separately for living participants as only few participants died in this study.
Time Frame: From randomization till death or end of study, whichever occurs first (Up to approximately 2.5 years)
Population: Safety population included all randomized participants classified according to the actual study treatment received, regardless of random assignment. Overall number of participants analyzed signifies participants who were alive.
Measure: Median (Full Range); unit: months
Arm/Group | Zevalin | Observation
Number analyzed (Participants) | 35 | 41
months | 8.90 [2.73 to 22.60] | 6.14 [0.07 to 21.32]

2. Primary Outcome: Overall Survival for Death
Description: OS was the time from randomization to death. OS for death calculated as (date of death - randomization date)+ 1/30.4375. Overall Survival was summarized separately for participants who were died as only few participants died in this study.
Time Frame: From randomization till death or end of study, whichever occurs first (Up to approximately 2.5 years)
Population: Safety population included all randomized participants classified according to the actual study treatment received, regardless of random assignment. Overall number of participants analyzed signifies participants who died.
Measure: Median (Full Range); unit: months
Arm/Group | Zevalin | Observation
Number analyzed (Participants) | 1 | 2
months | 16.76 [16.76 to 16.76] | 5.82 [1.94 to 9.69]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time interval between the date of randomization and the date of relapse or death from any cause.
Time Frame: From randomization till death or end of study, whichever occurs first (Up to approximately 2.5 years)
Population: Data for this outcome measure was not collected and analyzed due to early termination of study for sponsor business decision.
Arm/Group | Zevalin | Observation
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Survival Rate at 24 Months
Description: The OS rate at 24-month defined as the percentage of all randomized participants who died within 24 months of randomization.
Time Frame: 24 Months
Population: as for outcome 3
Arm/Group | Zevalin | Observation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose up to approximately 2.5 years
Description: Safety population included all randomized participants classified according to the actual study treatment received, regardless of random assignment.
Arm/Group | Zevalin | Observation
All-Cause Mortality (participants affected / at risk) | 1/36 | 2/43
Serious Adverse Events (participants affected / at risk) | 8/36 | 3/43
Other Adverse Events (participants affected / at risk) | 21/36 | 7/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zevalin (N=36) | Observation (N=43)
Neutropenia (Blood and lymphatic system disorders) | 4 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Death (General disorders) | 0 | 2
Lung infection (Infections and infestations) | 1 | 0
Platelet count decreased (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zevalin (N=36) | Observation (N=43)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 0
Constipation (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 10 | 2
Platelet count decreased (Investigations) | 6 | 0
Neutrophil count decreased (Investigations) | 6 | 0
White blood cell count decreased (Investigations) | 6 | 0
Lymphocyte count decreased (Investigations) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Headache (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to a sponsor business decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No